| PARTICIPANT INFORMATION SHEET |
|--------------------------------------------------------------|
| Screen to Save: A Colorectal Cancer Educational Intervention |
| NCT03907579 |
| Date: March 7, 2017 |

## DARTMOUTH COLLEGE/NORRIS COTTON CANCER CENTER

## Screen to Save

## RESEARCH PROJECT INFORMATION SHEET

Researchers at the Norris Cotton Cancer Center are conducting a research project called Screen to Save. The goal of this research is to understand if our colorectal cancer educational program helps improve people's understanding about colorectal cancer prevention and screening.

Your participation in this research is voluntary. The research involves three steps:

- 1. Complete a brief questionnaire that will take about 7 minutes to finish
- 2. Go through the colon with a tour guide and learn about colorectal cancer. That will take about 6 minutes
- 3. Complete another brief questionnaire that will take about 7 minutes

You may choose to not answer any or all questions. In all, we expect it will take about 20 minutes to complete this study. If you complete all three steps, you will be offered a \$10 gift card for your time.

Your answers on the questionnaires will be kept confidential. We won't even collect your name, contact information, or other identifying information.

Questions about the study should be directed to the researcher leading this study, Tracy Onega, PhD, MA, MS at (603) 653-3671, <u>Tracy.L.Onega@Dartmouth.edu</u>, or by mail at 1 Medical Center Drive, Hinman Box 7927, Lebanon, NH 03756. For general questions about research at Dartmouth, you should call the Office of the Committee for the Protection of Human Subjects at Dartmouth College (603) 646-6482.